CLINICAL TRIAL: NCT00652847
Title: Randomized Parallel Group Trial Of The Efficacy And Safety Of Ezetimibe With A Statin Versus Statin Dose Doubling In Patients With Persistent Primary Hypercholesterolemia
Brief Title: Randomized Parallel Group Trial Of The Efficacy And Safety Of Ezetimibe With A Statin Versus Statin Dose Doubling In Patients With Persistent Primary Hypercholesterolemia (0653-152)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0653-152; MK0653-152; 2008_005
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Hydroxymethylglutaryl-CoA Reductase Inhibitors

ARMS (2):
- group 1 (Experimental): group 1: ezetimibe 10 mg per day is added to actual statin regimen for 6 weeks followed by an observational phase of 6 months.
  Interventions: Drug: ezetimibe; Drug: statins
- Group 2 (Active Comparator): Group 2: patients on statins have their dose doubled for 6 weeks followed by another 6 month observational phase.
  Interventions: Drug: statins

INTERVENTIONS:
Drug: ezetimibe — ezetimibe 10 mg/day for a six week course of treatment.
  Other Names: Zetia®; MK0653
  Arms: group 1
Drug: statins — patients on statins have their dose doubled for 6 weeks followed by another 6 month observational phase

SUMMARY:
To compare the percent (%) change in plasma LDL-C concentration, after a six week course of treatment with ezetimibe 10 mg/day co-administered with an existing statin versus doubling of the existing statin dose

ELIGIBILITY:
Inclusion Criteria:

* Patients With A Diagnosis Of Primary Hypercholesterolemia And
* Who Are Defined As Being "High Risk" (10-Year Risk Of Coronary Artery Disease > 20 % Based On The Framingham Model Or History Of Diabetes Mellitus Or Any Atherosclerosis Disease)
* And Have Not Reached Their Recommended Ldl-C Target Levels Of 2.5 Mmol/L While On A Statin Alone

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1140 (Actual)
Dates: Start 2005-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The primary measure of efficacy will be the percent change in plasma LDL-cholesterol between baseline and the final study assessment after six weeks of treatment. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Shekhar Pandey A, Bissonnette S, Boukas S, Rampakakis E, Sampalis JS. Effectiveness and tolerability of ezetimibe co-administered with statins versus statin dose-doubling in high-risk patients with persistent hyperlipidemia: The EZE(STAT)2 trial. Arch Med Sci. 2011 Oct;7(5):767-75. doi: 10.5114/aoms.2011.25550. Epub 2011 Nov 8. PMID 22291820